CLINICAL TRIAL: NCT05231122
Title: Randomized Phase 2 Clinical Trial of Pembrolizumab Combined With Bevacizumab With or Without Agonist Anti-CD40 CDX-1140 in Patients With Recurrent Ovarian Cancer
Brief Title: Pembrolizumab Combined With Bevacizumab With or Without Agonist Anti-CD40 CDX-1140 for the Treatment of Patients With Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celldex Therapeutics (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I 1277721; NCI-2021-13609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 1277721 (Other: Roswell Park Cancer Institute); HT9425-23-1-1063 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-01-24; First posted 2022-02-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Clear Cell Adenocarcinoma; Platinum-Sensitive Ovarian Carcinoma; Recurrent Endometrial Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Fallopian Tube Endometrioid Adenocarcinoma; Recurrent Fallopian Tube Serous Adenocarcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian Serous Adenocarcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Primary Peritoneal Clear Cell Adenocarcinoma; Recurrent Primary Peritoneal Endometrioid Adenocarcinoma; Recurrent Primary Peritoneal Serous Adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; pembrolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (pembrolizumab, bevacizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes and bevacizumab IV over 30-90 minutes on day 1. Cycles repeat every 3 weeks until disease progression or development of unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (pembrolizumab, bevacizumab, CDX-1140) (Experimental): Patients receive pembrolizumab IV over 30 minutes, bevacizumab IV over 30-90 minutes, and CDX-1140 IV over 90 minutes on day 1. Cycles repeat every 3 weeks until disease progression or development of unacceptable toxicity.
  Interventions: Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140; Biological: Bevacizumab; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Anti-CD40 Agonist Monoclonal Antibody CDX-1140 — Given IV
  Other Names: Agonist CD40 Antibody CDX-1140; Anti-CD40 Agonistic Monoclonal Antibody CDX-1140; CDX 1140; CDX-1140
  Arms: Arm II (pembrolizumab, bevacizumab, CDX-1140)
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; Zirabev
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests whether pembrolizumab combined with bevacizumab with or without agonist anti-CD40 CDX-1140 works to shrink tumors in patients with ovarian cancer that has come back (recurrent). Anti-CD40 CDX-1140 works by stimulating certain immune cells within the tumor and, when combined with other immunotherapy treatments, may increase antitumor antibody production. Immunotherapy with monoclonal antibodies, such as pembrolizumab and bevacizumab, may help the body's immune system, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab and bevacizumab with anti-CD40 CDX-1140 may decrease symptoms, prolong survival, and improve quality of life in patients with ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of anti-CD40 agonist monoclonal antibody CDX-1140 (CDX-1140) combined with pembrolizumab and bevacizumab in patients with recurrent ovarian cancer (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).

II. Determine the objective response rate (ORR) per immune related response criteria (immune-modified Response Evaluation Criteria in Solid Tumors [iRECIST]).

SECONDARY OBJECTIVES:

I. Determine progression free survival (PFS), disease control rate (DCR) and overall survival (OS).

II. Changes in quality of life measures during the clinical trial (European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-Core 30 [QLQ-C30], EORTC QLQ-Ovarian Cancer Module [OV28] and Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF)].

EXPLORATORY OBJECTIVES:

I. Pharmacokinetic (PK)/anti-drug antibody (ADA) analysis for CDX-1140. II. Evaluate the immunologic and phenotypic changes in blood samples. III. To obtain data on changes in tumor microenvironment prior to and subsequent to therapy and, to screen for potential biomarkers to predict clinical benefit.

IV. Microbiome analysis from stool, tumor tissue.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pembrolizumab intravenously (IV) over 30 minutes and bevacizumab IV over 30-90 minutes on day 1. Cycles repeat every 3 weeks until disease progression or development of unacceptable toxicity.

ARM II: Patients receive pembrolizumab IV over 30 minutes, bevacizumab IV over 30-90 minutes, and CDX-1140 IV over 90 minutes on day 1. Cycles repeat every 3 weeks until disease progression or development of unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age.
* Recurrent serous (low grade or high grade), endometrioid, or clear cell recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer.
* Participant can be either platinum-sensitive or platinum-resistant, no more than 4 prior lines of treatment, and BRCA status must be known.

Neoadjuvant + adjuvant is considered one line.

* Participants may have received a prior PARPi, this will not be considered a separate line of therapy if received in maintenance.
* Participants may have received a prior anti-PD1/anti-PDL1 therapy or bevacizumab, these will not be considered a separate line of therapy.
* Any chemotherapy regimen change due to toxicity in the absence of disease progression will be considered part of the same line of therapy.
* Hormonal therapy for OC (e.g. Tamoxifen, aromatase inhibitors etc.) will not count as a separate line of prior therapy.

  * Anticipated lifespan greater than 6 months.
  * Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Patient has measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present.
  * All residual toxicity related to prior anti-cancer therapies (excluding alopecia, grade 2 fatigue, vitiligo, endocrinopathies on stable replacement therapy, grade 2 neuropathy from taxanes or platinum and grade 2 hearing loss from platinum) must be resolved to grade 1 severity or less (or returned to baseline) prior to receipt of study treatment.
  * Absolute neutrophil count (ANC): >= 1,500 /mcL.
  * Platelets: >= 100,000 / mcL.
  * Hemoglobin: >= 8 g/dL or 5.0 mmol/L transfusion allowed with adequate bone marrow function
  * Creatinine clearance >= 50 mL/min.
  * Urine protein creatinine ratio (UPCR) < 1 mg/dL prior to enrollment.
  * Total bilirubin: =< 2 X upper limit of normal (ULN) except patients with Gilbert's syndrome or liver involvement, who must have a total bilirubin =< 3 mg/dL.
  * Aspartate aminotransferase (AST) ( serum glutamic-oxaloacetic transaminase [SGOT] ) and alanine aminotransferase (ALT) ( serum glutamate pyruvate transaminase [SGPT]): =< 2.5 X ULN OR =< 5 X ULN for participants with liver metastases.
  * Albumin: > 2.5 mg/dL.
  * International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (APTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
  * Participant must be willing to undergo core or excisional biopsy of a tumor lesion within 7 days prior to the first dose of investigational product and after 3 cycles of treatment(prior to cycle 4-day 1: mandatory only if available) and, at the end of treatment (optional). Participants for whom newly obtained samples cannot be provided at baseline (e.g., inaccessible or subject safety concern), may submit an archived specimen, only upon agreement from the Prinicipal Investigator, if available).
  * A woman of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  * Participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication (participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year). Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
  * Participant (or legal representative) must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Primary platinum-refractory patients are excluded
* Has a nonepithelial cancer (germ cell tumors, sex cord-stromal tumors), borderline tumors, mucinous or seromucinous that is predominately mucinous, malignant Brenner's tumor, carcinosarcoma or undifferentiated carcinoma.
* Receipt of any antibody targeting T cell checkpoint or co-stimulation pathways within 4 weeks, use of any other monoclonal based therapies within 4 weeks, and all other immunotherapy (tumor vaccine, cytokine, or growth factor given to control the cancer) within 2 weeks prior to the planned start of study treatment.
* Has received prior systemic anticancer therapy (including investigational agents or maintenance therapy) within 28 days prior to the planned start of study treatment.

Hormonal therapy is allowed until the time of randomization

* Progression on prior immune checkpoint blockade therapy.
* Systemic radiation therapy within 4 weeks, prior focal radiotherapy within 2 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Major surgery within 4 weeks prior to the first dose of study treatment. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration and patients should be recovered.
* Known or prior malignancy requiring active treatment in the past 2 years. Exception: basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 3 years.
* Active, untreated central nervous system metastases. Patients with brain metastases identified at screening may be rescreened after the lesion(s) have been appropriately treated; patients with treated brain metastases should be neurologically stable for 4 weeks post-treatment and prior to study enrollment, and off corticosteroids for at least 2 weeks before administration of study drugs, and treated lesions should demonstrate no new growth on the re-screening scan.
* History of (non-infectious) pneumonitis or has current pneumonitis, including grade 1 (asymptomatic; clinical or diagnostic observations only; intervention not indicated) pneumonitis.
* History of severe hypersensitivity reactions to other monoclonal antibodies (mAbs).
* Prior therapy with any anti-CD40 antibody.
* Hypersensitivity to bevacizumab, pembrolizumab, or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid)
* Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months.
* Has an acute infection requiring systemic therapy
* Known immunodeficiency or active human immunodeficiency virus (HIV)
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA)and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Note: Hepatitis B and C screening tests are not required unless known history of HBV and HCV infection
* Has an active infection requiring systemic therapy
* Known immunodeficiency or active HIV
* Has received any investigational vaccines (i.e., those not licensed or approved for emergency use). Note: Any licensed COVID-19 vaccine (including for Emergency Use) is allowed in the study as long as they are mRNA vaccines, adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy.

Investigational vaccines (i.e., those not licensed or approved for Emergency Use) are not allowed.

* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Subject requires or is likely to require more than a two-week course of corticosteroids for intercurrent illness. Subject must complete the course of corticosteroids 2 weeks before screening to meet eligibility.
* Subject has a serious, non-healing wound, ulcer, or bone fracture.
* Subject has a clinically significant cardiovascular disease including:

  * Uncontrolled hypertension < 150/90 mmHg (may be rescreened after adequate control)
  * Myocardial infarction or unstable angina within 6 months prior to enrollment
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* New onset on thromboembolic event or hemorrhage within 6 weeks prior to randomization
* Subject has organ allografts.
* Subject has clinical symptoms or signs of partial or complete gastrointestinal obstruction or require parenteral hydration and/or nutrition.
* Pregnant or nursing female participants.
* Known active alcohol or drug abuse.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Evaluated according to National Cancer Institute Common Terminology Criteria for adverse events (NCI CTCAE) version (v)5.0. Will be summarized by cohort and grade using frequencies and relative frequencies.
Objective response rate (ORR) | Up to 2 years
  Will be summarized by cohort (with or without CDX 1140) using frequencies and relative frequencies, with the ORR estimated using 90% confidence intervals obtained by Jeffrey's prior method. The final analysis will be performed on all n=80 (40 in each cohort) evaluable patients; and if the p-value is less than or equal to 0.10, then the triplet regimen will be considered superior with respect to response.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From first day of treatment until disease progression or date of death from any cause, assessed up to 2 years
  Will be summarized by cohort using standard Kaplan-Meier methods, with estimates of the median obtained with 90% confidence intervals. PFS will be compared between cohorts using a one-sided log-rank test.
Overall survival (OS) | From first day of treatment until disease progression or date of death from any cause, assessed up to 2 years
  Will be summarized by cohort using standard Kaplan-Meier methods, with estimates of the median obtained with 90% confidence intervals. OS will be compared between cohorts using a one-sided log-rank test.
Disease control rate (DCR) | Up to 2 years
  Will be summarized by cohort using frequencies and relative frequencies, with the DCR estimated by cohort using 90% confidence intervals obtained by Jeffrey's prior method. The DCR will be compared between cohorts using a one-sided Cohran-Mantel-Haenszel test.
Quality of Life (QoL)EORTC QLQ-C30 | Up to 2 years
  European Organization for Research and Treatment of Cancer (EORTC) QLQ-30 consists of 28 questions with answers that range from 1 (Not At All) to 4 (Very Much) and 2 questions that range from 1 (Very Poor) to 7 (Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - M D Anderson Cancer Center, Houston, Texas